CLINICAL TRIAL: NCT04707196
Title: A Single-Arm, Phase 4 Study of Abemaciclib, a CDK4 and CDK6 Inhibitor, in Combination With Endocrine Therapy (Anastrozole/Letrozole or Fulvestrant) in Participants With Hormone Receptor Positive, Human Epidermal Growth Factor Receptor 2 Negative Locally Advanced and/or Metastatic Breast Cancer in India
Brief Title: A Study of Abemaciclib in Indian Women With Advanced Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17782; I3Y-IN-JPEC (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — abemaciclib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Abemaciclib + NSAI or Fulvestrant (Experimental): Participants received abemaciclib 150 milligram (mg) orally twice daily, on days 1 through 28 of a 28-day cycle, for up to 6 cycles or less in case of disease progression, or any other discontinuation criterion is met, plus either NSAI (nonsteroidal aromatase inhibitors - anastrozole or letrozole) administered orally as per standard of care or fulvestrant administered intramuscularly as per standard of care.
  Interventions: Drug: Abemaciclib; Drug: Nonsteroidal Aromatase Inhibitor (NSAI); Drug: Fulvestrant

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
Drug: Nonsteroidal Aromatase Inhibitor (NSAI) — Letrozole or anastrozole administered orally (physician choice)
Drug: Fulvestrant — Administered intramuscularly

SUMMARY:
The main purpose of this study is to learn more about the safety and tolerability of abemaciclib when given in combination with hormone therapy in Indian women with advanced breast cancer. Participants must have hormone receptor positive (HR+), human epidermal growth factor receptor 2 negative (HER2-) breast cancer and must live in India. For each participant, the study could last up to eight months and may include up to eight visits to the study center.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of hormone receptor-positive (HR+), human epidermal growth factor receptor 2-negative (HER2-) breast cancer
* Have locoregionally recurrent disease not amenable to resection or radiation therapy with curative intent or metastatic disease
* Have postmenopausal status
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have adequate organ function
* Have discontinued previous cytotoxic therapies, biological agents, investigational agents, and radiotherapy
* Are able to swallow oral formulation

Exclusion Criteria:

* Have visceral crisis, lymphangitic spread, or leptomeningeal carcinomatosis.
* Have clinical evidence or history of central nervous system metastasis.
* Have received prior treatment with chemotherapy (except for neoadjuvant/adjuvant chemotherapy), fulvestrant, everolimus, or any cyclin-dependent kinase (CDK) 4 & 6 inhibitor.
* Have received recent (within 28 days prior to study intervention) live vaccination (for example, yellow fever). Seasonal flu vaccinations that do not contain a live virus are permitted.
* Have a personal history of presyncope or syncope of either unexplained or cardiovascular etiology, ventricular tachycardia, ventricular fibrillation, or sudden cardiac arrest.
* Have inflammatory breast cancer or a history of any other cancer (except nonmelanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission with no therapy for a minimum of 3 years.
* Have received an autologous or allogeneic stem-cell transplant
* Have clinically relevant active bacterial or fungal infection, or detectable viral infection (for example, human immunodeficiency virus or viral hepatitis). Screening is not required for enrolment.
* Are pregnant or breastfeeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- India (15):
  - MNJ Institute of Oncology, Hyderabad, Andhra Pradesh
  - Indira Gandhi Institute of Medical Sciences, Patna, Bihar
  - Nirmal Hospital Pvt Ltd., Surat, Gujarat
  - Unique Hospital Multispecialty & Research Institute, Surat, Gujarat
  - Kailash Cancer Hospital & Research Centre (KCHRC), Waghodia, Gujarat
  - HCG Cancer Centre, Kalinga Rao Road, Bengaluru, Karnataka
  - Regional Cancer Centre, Trivandrum, Kerala
  - SRJ-CBCC Cancer Hospital, Indore, Madhya Pradesh
  - Kingsway Hospital, Nagpur, Maharashtra
  - Meditrina Institute of Medical Sciences, Nagpur, Maharashtra
  - HCG Manavata Cancer Centre, Nashik, Maharashtra
  - Ruby Hall Clinic and Grant Medical Foundation, Pune, Maharashtra
  - Rajiv Gandhi Cancer Institute And Research Centre, New Delhi, National Capital Territory of Delhi
  - Apollo Gleneagles Hospitals Kolkata, Kolkata, West Bengal
  - Max Superspeciality Hospital, Chandigarh

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Abemaciclib + NSAI: Participants received abemaciclib 150 milligram (mg) orally twice daily, on days 1 through 28 of a 28-day cycle, for up to 6 cycles or less in case of disease progression, or any other discontinuation criterion is met, plus NSAI (nonsteroidal aromatase inhibitors - either anastrozole or letrozole) administered orally as per standard of care.
- Abemaciclib + Fulvestrant: Participants received abemaciclib 150 mg orally twice daily, on days 1 through 28 of a 28-day cycle, for up to 6 cycles or less in case of disease progression, or any other discontinuation criterion is met, plus fulvestrant administered intramuscularly as per standard of care.
Period: Overall Study
Arm/Group | Abemaciclib + NSAI | Abemaciclib + Fulvestrant
Started | 137 | 63
Received at Least 1 Dose of Study Drug | 137 | 63
Completed (Participants who completed 6 cycles of study intervention were considered completers.) | 108 | 43
Not Completed | 29 | 20
Not completed — Withdrawal by Subject | 9 | 6
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 4 | 1
Not completed — Adverse Event | 2 | 2
Not completed — Death | 3 | 1
Not completed — Non-compliance with study drug | 1 | 0
Not completed — Progressive disease | 9 | 10

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Abemaciclib + NSAI: Participants received abemaciclib 150 mg orally twice daily, on days 1 through 28 of a 28-day cycle, for up to 6 cycles or less in case of disease progression, or any other discontinuation criterion is met, plus NSAI (nonsteroidal aromatase inhibitors - either anastrozole or letrozole) administered orally as per standard of care.
- Total: Total of all reporting groups
Arm/Group | Abemaciclib + NSAI | Abemaciclib + Fulvestrant | Total
Number analyzed (Participants) | 137 | 63 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.60 (11.66) | 51.80 (12.54) | 54.40 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 63 | 200
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 137 | 63 | 200
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  India | 137 | 63 | 200

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing at Least One Treatment-Emergent Adverse Event
Description: Treatment-emergent adverse events (TEAEs) are defined as any adverse events that started at the time of, or after the, first study medication administration as well as those events that started prior to the first study drug administration, but which worsened after the first study medication administration. The reported data reflects the unique percentage of participants who experienced any serious and other non-serious adverse events. A summary of serious and other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline until end of follow-up (Up To 7 Months)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Abemaciclib + NSAI | Abemaciclib + Fulvestrant
Number analyzed (Participants) | 137 | 63
percentage of participants | 78.1 | 69.8

2. Secondary Outcome: Percentage of Participants Who Discontinued From Study Treatment Due to Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Baseline until end of study treatment (Up To 6 Months)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Abemaciclib + NSAI | Abemaciclib + Fulvestrant
Number analyzed (Participants) | 137 | 63
percentage of participants | 3.6 | 4.8

ADVERSE EVENTS:
Time Frame: Baseline until end of follow-up (Up To 7 Months)
Description: All participants who received at least one dose of study drug.
Arm/Group | Abemaciclib + NSAI | Abemaciclib + Fulvestrant
All-Cause Mortality (participants affected / at risk) | 3/137 | 1/63
Serious Adverse Events (participants affected / at risk) | 9/137 | 5/63
Other Adverse Events (participants affected / at risk) | 105/137 | 44/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib + NSAI (N=137) | Abemaciclib + Fulvestrant (N=63)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (2)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib + NSAI (N=137) | Abemaciclib + Fulvestrant (N=63)
Anaemia (Blood and lymphatic system disorders) | 32 (48) | 14 (22)
Leukopenia (Blood and lymphatic system disorders) | 19 (39) | 6 (13)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 34 (61) | 11 (22)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (7) | 4 (16)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Central serous chorioretinopathy (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 11 (20) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 41 (132) | 18 (41)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (3) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperchlorhydria (Gastrointestinal disorders) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (21) | 10 (10)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 4 (5)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 17 (27) | 13 (23)
Asthenia (General disorders) | 7 (11) | 3 (4)
Fatigue (General disorders) | 8 (13) | 13 (21)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 4 (4)
Pain (General disorders) | 2 (2) | 1 (1)
Peripheral swelling (General disorders) | 3 (3) | 2 (3)
Pyrexia (General disorders) | 7 (8) | 6 (6)
Swelling face (General disorders) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 3 (3) | 4 (4)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1)
Tinea infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 2 (3)
Blood creatine increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 10 (15) | 2 (3)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
Cystatin c increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (4)
Neutrophil count decreased (Investigations) | 6 (10) | 9 (13)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Vitamin b12 decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 6 (7) | 7 (8)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 5 (6)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (5) | 3 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (11) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 4 (6)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 3 (3)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT04707196/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT04707196/SAP_001.pdf